CLINICAL TRIAL: NCT01301170
Title: The Effectiveness of Dry Needling for Patients With Neck Pain: A Randomized Clinical Trial
Brief Title: Study Evaluating the Benefit of Dry Needling for Patients With Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Integrated Therapy Practice PC (Other)
Responsible Party: Rob Sillevis, Integrated Therapy Practice PC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UR-0922-129
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Neck Pain
Keywords: Neck pain; Dry Needling; Manual Therapy; Manipulation
MeSH Terms: conditions — Neck Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: dry needling — The needling will take place bilaterally at both the suboccipital region and the paravertebral muscles between C4 and T4. The needling will take place with the patient in the prone position. Following all needle placement, they will rotated clockwise till the point that tension on the needle is felt by the therapist. This will create more tension between the needle and tissue fibers, after which the needles were removed.

SUMMARY:
The purpose of this study is to determine whether individuals with neck pain will respond favorably to a program of manual therapy, directed at the cervical and thoracic spine (including thrust manipulation), and exercise, in combination with dry needling, as compared to manual therapy, directed to the cervical and thoracic spine (including thrust manipulation), and an exercise program alone.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-60 years old
2. Primary complaint of neck pain
3. Restricted cervical extension/and or cervical rotation ROM
4. Neck Disability Index > 20 points

Exclusion Criteria:

1. Red flags noted in the patient's Neck Medical Screening Questionnaire (i.e. tumor, fracture, metabolic diseases, RA, osteoporosis, prolonged history of steroid use, symptoms of vertebrobasilary insufficiency, pregnancy, cervical spinal stenosis, bilateral upper extremity symptoms etc.
2. Use of blood thinners
3. History of whiplash injury within the past six weeks
4. Evidence of central nervous system involvement, to include hyperreflexia, sensory disturbances in the hand, intrinsic muscle wasting of the hands, unsteadiness during walking, nystagmus, loss of visual acuity, impaired sensation of the face, altered taste, the presence of pathological reflexes (i.e. positive Hoffman's and/or Babinski reflexes), etc.
5. Two or more positive neurologic signs consistent with nerve root compression, including any two of the following:

   * Muscle weakness involving a major muscle group of the upper extremity
   * Diminished upper extremity muscle stretch reflex (biceps brachii, brachioradialis, or triceps)
   * Diminished or absent sensation to pinprick in any upper extremity dermatome
6. Prior surgery to the neck or thoracic spine
7. Chiropractic, Physical Therapy, or Acupuncture treatment for their neck pain in the last 12-months
8. Workers compensation or pending legal action regarding their headaches
9. Insufficient English language skills to complete all questionnaires
10. Inability to comply with treatment and follow-up schedule

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-11 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
neck disability index (NDI) | 4,12, 24 weeks

SECONDARY OUTCOMES:
Patient Global Rating of Change (GROC) | 4, 12, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rob Sillevis, PT,DPT,PhD, Principal Investigator — adjunct faculty University of St. Augustine for Health Sciences
Locations (1):
- Integrated Therapy Practice PC, Hobart, Indiana, United States